CLINICAL TRIAL: NCT07089641
Title: A Phase Ib Open Label Clinical Trial to Evaluate the Safety and Efficacy of ERAS-801 in Surgically Accessible Recurrent Glioblastoma Patients With EGFR Amplification or Mutation (ERAS801-SARG)
Brief Title: ERAS-801 for the Treatment of Resectable and Progressive or Recurrent IDH Wildtype Grade IV Glioblastoma or Astrocytoma With an EGFR Amplification or Mutation, ERAS801-SARG Trial
Acronym: ERAS801-SARG
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-5945; NCI-2025-00605 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-04-10; First posted 2025-07-28 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-07

CONDITIONS: IDH Wildtype Glioblastoma; Recurrent Astrocytoma; IDH Wildtype Recurrent Glioblastoma; Resectable Astrocytoma; Resectable Glioblastoma
MeSH Terms: conditions — Astrocytoma | interventions — Specimen Handling; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (ERAS-801) (Experimental): Patients receive ERAS-801 PO QD for 8-14 days prior to undergoing scheduled surgical resection. Starting no more than 28 days after surgery, patients then receive ERAS-801 PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo ECHO, urine and blood sample collection and brain MRI throughout the study. Additionally, patients undergo CSF sample collection at the time of surgery and FDG PET on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Echocardiography Test; Drug: EGFR Inhibitor ERAS-801; Other: Fludeoxyglucose F-18; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Surgical Procedure

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo urine, blood, and CSF sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: EGFR Inhibitor ERAS-801 — Given PO
  Other Names: ERAS 801; ERAS-801; ERAS801
Other: Fludeoxyglucose F-18 — Given FDG
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Procedure: Magnetic Resonance Imaging — Undergo brain MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo FDG PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Surgical Procedure — Undergo surgical resection
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery

SUMMARY:
This phase Ib trial tests the safety and side effects of ERAS-801 in treating patients with isocitrate dehydrogenase (IDH) wildtype, epidermal growth factor receptor (EGFR) amplified or mutated grade IV glioblastoma or astrocytoma that can be removed by surgery (resectable) and that is growing, spreading, or getting worse (progressive) or that has come back after a period of improvement (recurrent). Glioblastoma is the most common brain cancer in adults and survival rates remain poor despite treatment including surgery, radiation and chemotherapy. EGFR is a protein found on the surface of some cells, to which epidermal growth factor binds, causing the cells to divide. It is found at abnormally high levels on the surface of many types of tumor cells, so these cells may divide excessively in the presence of epidermal growth factor. ERAS-801, an EGFR inhibitor that can penetrate the central nervous system, binds to the tumor cells that express EGFR and may help shrink or slow the growth of the tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the glucose utilization in the tumor from the glioblastoma patients treated with EGFR inhibitor ERAS-801 (ERAS-801).

II. To evaluate the influence of ERAS-801 treatment on the apoptotic machinery in recurrent glioblastoma.

III. To evaluate the safety and tolerability of ERAS-801 recommended phase 2 dose (RP2D) in recurrent glioblastoma.

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetic (PK) profile in plasma, cerebrospinal fluid (CSF), and tumor tissue of ERAS-801 in recurrent glioblastomas.

II. To evaluate the pharmacodynamic (PD) impact of ERAS-801 treatment in recurrent glioblastomas.

III. To evaluate whether glycolytic index (GI) measured by fludeoxyglucose F-18 (FDG)-positron emission tomography (PET) and metabolic magnetic resonance imaging (MRI) correlates with clinical responses in recurrent glioblastomas treated with ERAS-801.

IV. To evaluate whether potential of hydrogen (pH)-weighted chemical exchange saturation transfer (CEST)-spin-and-gradient echo (SAGE)-echoplanar imaging (EPI) contrast measured by metabolic MRI correlates with clinical responses in recurrent glioblastomas treated with ERAS-801.

EXPLORATORY OBJECTIVES:

I. To evaluate the associations between exploratory biomarkers, clinical outcomes, and adverse events which include:

Ia. Estimating the efficacy of ERAS-801 through 6 month progression free survival (PFS6), progression free survival (PFS), and overall survival (OS) as defined by modified Response Assessment in Neuro-Oncology criteria (mRANO)/Response Assessment in Neuro-Oncology criteria (RANO) 2.0; Ib. Exploring whether glycolytic index (GI) and pH-weighted CEST-SAGE-EPI contrast correlates with clinical responses; Ic. Exploring whether there are alterations of key glycolytic enzymes and/or other transcriptional changes linked to EGFR occur with ERAS-801 treatment; Id. Exploring whether there are changes in percent of tumor cells that have immunohistochemical positive staining for the KI67 antigen after ERAS-801 treatment; Ie. Exploring the associations between the various biomarker evaluations (tissue and imaging), clinical outcome measures and adverse events.

OUTLINE:

Patients receive ERAS-801 orally (PO) once daily (QD) for 8-14 days prior to undergoing scheduled surgical resection. Starting no more than 28 days after surgery, patients then receive ERAS-801 PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo echocardiography (ECHO), urine and blood sample collection and brain MRI throughout the study. Additionally, patients undergo CSF sample collection at the time of surgery and FDG PET on study.

After completion of study treatment, patients are followed up at 30 days, then every 2 months up to documented disease progression, death, or the end of the study. Patients with disease progression are followed up every 12 weeks up to death, withdrawal of consent, or the end of the trial, whichever, occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older on the day of signing informed consent
* Patients must have histologically proven surgically accessible World Health Organization (WHO) grade IV glioblastoma/astrocytoma, which is progressive or recurrent following radiation therapy +/- chemotherapy
* Patient tumor sample must have wild type IDH with evidence of EGFR mutation/amplification by Clinical Laboratory Improvement Act (CLIA)-certified laboratory assay
* Patients may have had no more than two prior recurrences
* Patient must be able to tolerate MRIs. Pre-study enrollment MRIs must be available for central review, including at least the immediate pre-progression scan and the scan demonstrating progression. Patients must have measurable, by RANO, supratentorial contrast-enhancing progressive or recurrent high-grade glioma by MRI imaging within 7 days of starting treatment
* Patients must have recovered from severe toxicity of prior therapy. The following intervals from previous treatments are required to be eligible:

  * 12 weeks from the completion of radiation
  * 6 weeks from a nitrosourea chemotherapy
  * 3 weeks from a non-nitrosourea chemotherapy
  * 4 weeks from any investigational (not Food and Drug Administration [FDA]-approved) agents
  * 4 weeks from the last treatment with bevacizumab
  * 2 weeks from administration of a non-cytotoxic, FDA-approved agent other than bevacizumab (e.g., hydroxychloroquine, etc.)
  * 1 week from the tumor treating fields
* Patients must be undergoing surgery that is clinically indicated as determined by their care providers. Patients must be eligible for surgical resection according to the following criteria:

  * Expectation that the surgeon can resect at least 500 mg of tumor from enhancing tumor and 100 mg from non-enhancing tumor with low risk of inducing neurological injury
* Paraffin embedded tissue must be available from initial surgical resection at diagnosis (prior to any treatment). The following amount of tissue is requested: 1 formalin-fixed, paraffin embedded (FFPE) tissue block (preferred) or 30 FFPE unstained slides (5µm thick)
* Patients must have a Karnofsky performance status ≥ 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
* Absolute neutrophil count (ANC) ≥ 1000/uL
* Platelets ≥ 100,000/uL
* Hemoglobin ≥ 9.0 g/dL or ≥ 5.6 mmol/L

  * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks
* Creatinine ≤ 1 x upper limit of normal (ULN) OR measured or calculated creatinine clearance ≥ 30 mL/min for participant with creatinine levels > 1 x institutional ULN (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl])

  * Creatinine clearance (CrCl) should be calculated per institutional standard
* Total bilirubin ≤ 1.5 x ULN unless with Gilbert's syndrome
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x ULN
* International normalized ratio (INR) OR prothrombin time (PT) activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
* Patients must have left ventricular ejection fraction (LVEF) within normal institutional limits within 21 days of starting treatment
* Patients must have a 12-lead electrocardiogram performed within 2 weeks of treatment start with Fridericia's formula-corrected QT interval (QTcF) < 450 msec
* Patients must be able to provide written informed consent
* Women of childbearing potential must have a negative urine or serum pregnancy test 7 days prior to the first dose
* Women of childbearing potential and men must agree to use adequate method of contraception for the duration of study participation and for 30 days after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 4 months after the last dose of study drug
* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder. Patients with prior malignancies must be disease-free for > three years
* Patients must be able to swallow medication by mouth

Exclusion Criteria:

* Participants may not be receiving any other investigational agents
* Participants with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to ERAS-801 are ineligible
* Participants with prior therapy with EGFR inhibitors are ineligible because treatment with EGFR kinase inhibitors or other EGFR-targeted agents has the potential to deplete the tumor of EGFR-amplified or EGFR mutant cell populations and confound the evaluation of ERAS-801 effects on participants
* Participants on enzyme-inducing anti-epileptic drugs (EIAED) are not eligible for treatment on this protocol. Patients may be on non-enzyme inducing anti-epileptic drugs or not be taking any anti-epileptic drugs. Patients previously treated with EIAED may be enrolled if they have been off the EIAED for 10 days or more prior to the first dose of ERAS-801
* Participants must not have evidence of significant hematologic, renal, or hepatic dysfunction
* Participants must not have evidence of significant intracranial hemorrhage
* Participants with clinically significant cardiovascular disease including, but not limited to:

  * Myocardial infarction or unstable angina within the 6 months prior to the first dose of study drug
  * Clinically significant cardiac arrhythmia
  * Prolonged QTcF > 450 ms
  * Uncontrolled (persistent) hypertension: systolic blood pressure > 180 mmHg; diastolic blood pressure > 100 mmHg
  * Congestive heart failure (New York Heart Association class III-IV)
  * Use of pacemaker
  * Pulmonary embolism < 30 days
* Participants with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible
* Pregnant women are excluded from this study because ERAS-801 has unknown potential for teratogenic or abortifacients effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ERAS-801, breastfeeding should be discontinued if the mother is treated with ERAS-801
* Participants currently using or anticipating need to use drugs, food, or herbal supplements known to be strong or moderate inducers or inhibitors of CYP3A4, CYP2C8, and/or CYP2D6 and P-glycoprotein (P-gp) substrates within 10 days of study enrollment are ineligible
* Participants who have acute or currently active/requiring anti-viral therapy hepatic or biliary disease are ineligible (with the exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases from the primary brain tumor, or stable chronic liver disease per investigator assessment)
* Patients with gastrointestinal conditions that may affect reliable administration/absorption of medications including difficulty swallowing/unable to swallow pills; malabsorption syndrome; refractory nausea and vomiting, chronic gastrointestinal (GI) disease or previous significant bowel resection with clinically significant sequelae are ineligible
* Participants receiving P-gp inhibitors are ineligible
* Patients who have known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | From enrollment to 30 days after the last dose of study treatment
  Adverse events will be described by the National Cancer Institute Common Terminology Criteria for Adverse Events version 5. Will be presented using a 95% confidence interval and 2-sided p-value, combined with Bayesian posterior means and High Posterior Density intervals. Descriptive summaries and data visualization will be used
Fludeoxyglucose F-18 (FDG) tumor uptake | Time Frame (Day 1 to Day 8 during pre-surgery treatment);at Baseline prior to Day 1 of pre-surgery study treatment & on Day 8 of Pre-surgery study treatment
  FDG positron emission tomography (PET), as measured by median normalized FDG standardized uptake value (SUV) within the contrast enhancing tumor, will be compared to estimate the change in FDG uptake in the tumor. A formal test for the mean difference will be based on a paired T-test. 95% confidence intervals will be used to quantify uncertainty in estimation

SECONDARY OUTCOMES:
Change in glycolytic index (GI) | Time Frame ( Day 1 to Day 8 during pre-surgery treatment); at Baseline prior to Day 1 of pre-surgery study treatment & on Day 8 of Pre-surgery study treatment
  The GI measurement will be measured by the product of FDG PET SUV and potential of hydrogen (pH)-weighted chemical exchange saturation transfer (CEST)-spin-and-gradient echo (SAGE)- echoplanar imaging (EPI) and will be compared to estimate the change in GI in the tumor area as a surrogate for changes in glycolytic flux.
pH-weighted CEST-SAGE-EPI | Time Frame ( Day 1 to Day 8 during pre-surgery treatment); at Baseline prior to Day 1 of pre-surgery study treatment & on Day 8 of Pre-surgery study treatment
  Amine proton CEST-SAGE-EPI will be evaluated for change in acidity in the tumor. Continued monitoring for tumor acidity will occur throughout the study treatment cycles.
Level of ERAS-801 | Pre-surgery: Day 1, day 8, day 9; post-surgery: day 1 of each cycle (28 day cycle)
  Blood, cerebrospinal fluid (CSF) and frozen tumor tissue will be collected to investigate the level of ERAS-801. Serial blood samples for determination of study drug and its metabolites in plasma will be taken at pre-dose on Day 1 of pre-surgery study treatment, on Day 8 of Pre-surgery study treatment, at the time of surgery and then at the beginning of each post-surgery treatment cycle (every 28 days). CSF will be collected at the time of surgery. Frozen tumor samples from the protocol on-study surgery will be collected at the time of the protocol surgery. Blood samples will be used to determine the drug concentration in the plasma. Any residual back-up samples may be used for additional exploratory biomarker research.

CONTACTS AND LOCATIONS:
Overall Officials: Phioanh Nghiemphu, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States